CLINICAL TRIAL: NCT05188989
Title: A Multi-Center ,Randomized, Double-Blind, Placebo-Controlled, Study to Evaluate the Efficacy and Safety of TPN171H in Patients With Erectile Dysfunction
Brief Title: Efficacy and Safety Study of TPN171H Tablets in Erectile Dysfunction.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TPN171H-E301
Record Dates: First submitted 2021-12-29; First posted 2022-01-12 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TPN171H 2.5mg group (Experimental)
  Interventions: Drug: TPN171H 2.5mg group
- TPN171H 5mg group (Experimental)
  Interventions: Drug: TPN171H 5mg group
- TPN171H 10mg group (Experimental)
  Interventions: Drug: TPN171H 10mg group
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo group

INTERVENTIONS:
Drug: TPN171H 2.5mg group — TPN171H 2.5mg taken orally on demand 0.5-4 hour prior to sexual intercourse
  Other Names: Simmerafil
  Arms: TPN171H 2.5mg group
Drug: TPN171H 5mg group — TPN171H 5mg taken orally on demand 0.5-4 hour prior to sexual intercourse
  Other Names: Simmerafil
  Arms: TPN171H 5mg group
Drug: TPN171H 10mg group — TPN171H 10mg taken orally on demand 0.5-4 hour prior to sexual intercourse
  Other Names: Simmerafil
  Arms: TPN171H 10mg group
Drug: Placebo group — Placebo taken orally on demand 0.5-4 hour prior to sexual intercourse
  Arms: Placebo group

SUMMARY:
This is a multicenter, randomized, double blind, placebo-controlled, parallel design study to evaluate the efficacy and safety of TPN171H in men with erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 65 years (inclusive)
* Males with ED at least 6 months
* IIEF-5 ≤ 21 at visit 1
* Patients in a stable, heterosexual relationship for at least 3 months and during the study;
* Patients who are willing to stay away from any other medicines or treatments for ED during this study period
* Patients who are willing to have 4 or more attempts of sexual intercourse per 4 weeks, demonstrated compliance with the study protocol, including drug administration, diary completion, and scheduled study visits, during the qualifying trial;
* Patients who are willing to take proper contraceptive during the study and within 3 months after the study completed;
* At the end of the untreated baseline period, the following conditions are met：（1）The subject must make at least four attempts at sexual intercourse during the untreated baseline period. （2）At least 50% of attempts during this period must be unsuccessful,（unsuccess means at least one of the first three questions should be answered "No" in SEP）.（3）5≤IIEF-EF≤25.
* Patients who have voluntarily decided to participate in this study, and signed the informed consent form.

Exclusion Criteria:

* Patients who have a history of hypersensitivity to other PDE5 inhibitors or TPN171H;
* Patients with anatomical malformations of the penis;
* Patients with primary hypoactive sexual desire;
* Patients with ED, which is caused by any other primary sexual disorder
* Patients with ED ,which is caused by spinal injury or have had a radical prostatectomy or other surgery
* Patients who have a penile implant
* Patients who have not responded to PDE5 inhibitors or who have an adverse reaction leading to discontinuation
* CYP3A4 potent inhibitors, potent inducers, and moderate inducers (except topical drugs) should be used within 28 days before the start of treatment or during the trial period.
* Subjects who are taking nitrate or NO donor drugs, anti-androgens, guanylate cyclase agonists, or other drugs or treatments for the treatment of ED and cannot be discontinued
* Patients with the following cardiovascular disease:
* Myocardial infarction or stroke within the last 6 months; Unstable angina or angina occurring during sexual intercourse; New York Heart Association Class 2 or greater heart failure in the last 6 months; Uncontrolled hypotension (<90/60mmHg), uncontrolled hypertension (≥160/95mmHg); Orthostatic hypotension.
* Diabetic patients whose FBS is over 1.5 fold of normal value, or whose HbA1c >9%, or with diabetes complications, such as diabetic nephropathy, peripheral neuropathy;
* Patients with hepatic or renal dysfunction as per the following: AST, ALT>2*ULN, serum creatinine exceeds 20% of the upper limit of normal value;
* Patients with active gastrointestinal ulcers and bleeding disorders;
* Patients who have a history of NAION, or with a known genetically degenerative retinopathy, including retinitis pigmentosa;
* Patients who have a history of sudden decrease or loss of hearing;
* Patients with a history of severe central nervous system injury or peripheral muscular neurological disease in the past 6 months.
* Patient with a history of malignancy;
* Patients with significant neurological abnormalities;
* Patients with alcohol addiction
* Patients with persistent abuse of drugs of dependence;
* Patients who are planning to father a baby or are in a relationship with a pregnant partner.
* Patients who have a childbirth plan during the trial period and within 3 months after the trial.
* Patients who are participating in the past 3 months from any other clinical trial
* For other reasons besides the aforementioned cases, patient whose participation is deemed inappropriate due to clinically significant findings according to the medical decision of the principal investigator or the study personnel.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 765 (Actual)
Dates: Start 2021-12-31 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in the International Index of Erectile Function - Erectile Function Domain (IIEF-EF) at Week 12 | baseline and 12 weeks
  The primary efficacy variable was the change in the EF domain scores of the IIEF questionnaire from baseline, calculated by comparing total scores from questions 1-5 and 15 from the IIEF questionnaire .
Change From Baseline in Question 2 of the Patient Sexual Encounter Profile (SEP) Diary at Week 12 in Percentage of Yes Responses | baseline and 12 weeks
  Assessed was the mean change from baseline in the percentage of Yes responses to the SEP diary Question 2. "Were you able to insert your penis into your partner's vagina when you are trying to have sex ?" Data are presented as the mean percentage of yes responses per participant.
Change From Baseline in Question 3 of the Patient Sexual Encounter Profile (SEP) Diary at Week 12 in Percentage of Yes Responses | baseline and 12 weeks
  Assessed was the mean change from baseline in the percentage of Yes responses to the SEP diary Question 3. "Did your erection last long enough for you to have successful intercourse?" Data are presented as the mean percentage of yes responses per participant.

SECONDARY OUTCOMES:
Change From Baseline in the International Index of Erectile Function - Erectile Function Domain (IIEF-EF) at Week 4、8 | baseline ,4 weeks and 8 weeks
  The primary efficacy variable was the change in the EF domain scores of the IIEF questionnaire from baseline, calculated by comparing total scores from questions 1-5 and 15 from the IIEF questionnaire .
Change From Baseline in the International Index of Erectile Function - Erectile Function Domain (IIEF-EF) ≥26 at Week 4、8、12 | baseline , 4 weeks , 8 weeks ,12 weeks
  Assessed was the changes in the number of subjects whose IIEF domain score at the 8th week visit was ≥26.
Change From Baseline to 4 Week , 8 Week and 12 Week Endpoint in International Index of Erectile Function (IIEF),Orgasmic Functions,Sexual Desire,Intercourse Satisfaction, Overall Satisfaction | baseline , 4 weeks , 8 weeks ,12 weeks
  Self-reported ,Orgasmic Functions,Sexual Desire,Intercourse Satisfaction, Overall Satisfaction over the past 12 weeks.
Change From Baseline in Question 2 of the Patient Sexual Encounter Profile (SEP) Diary at Week 4 in Percentage of Yes Responses | baseline , 4 weeks , 8 weeks
  Assessed was the mean change from baseline in the percentage of Yes responses to the SEP diary Question 2. "Were you able to insert your penis into your partner's vagina when you are trying to have sex?" Data are presented as the mean percentage of yes responses per participant.
Sexual Encounter Profile (SEP) Diary, Question 3 Change From Baseline to Week 4 in Percentage of Yes Responses | baseline , 4 weeks , 8 weeks
  Assessed was the mean change from baseline in the percentage of Yes responses to the SEP diary Question 3. "Did your erection last long enough for you to have successful intercourse?" Data are presented as the mean percentage of yes responses per participant.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Jiang, Principal Investigator — Peking University Third Hospital
Locations (49):
- China (49):
  - The Second People's Hospital of Hefei, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - The first affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Xiyuan Hospital china Academy of chinese Medical Sciences, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Shenzhen University General Hospital, Shenzhen, Guangdong
  - Songgang People's Hospital, Shenzhen, Guangdong
  - The Eighth Affiliated Hospital Sun Yat-sen University, Shenzhen, Guangdong
  - Zhuhai People's Hospital, Zhuhai, Guangdong
  - Liuzhou peopleˊs Hospital, Liuchow, Guangxi
  - The Second Nanning People's Hospital, Nanning, Guangxi
  - The First Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - People's Hospital of zhengzhou, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhenzhou, Henan
  - Tongji Medical College of HUST, Wuhan, Hubei
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Provincial Hospital of Chinese Medicine, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Nanchang reproductive hospital, Nanchang, Jiangxi
  - First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Affiliated Hospital to Changchun University of Traditional Medicine, Changchun, Jilin
  - The Frist Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Qinghai university affiliated hospital, Xining, Qinghai
  - Shandong Provincial Hospital, Jinan, Shandong
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Shanghai Ceneral Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pudong Hospital ,Fudan university PuDong Medical center, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Sichuan Academy of Medical Sciences.Sichuan Provincial People's Hospital, Chengdou, Sichuan
  - Clinical Medical College & Affiliated Hospital of Chengdu University, Chengdou, Sichuan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No